CLINICAL TRIAL: NCT06699316
Title: Individualized Prognostic Counseling on Life Expectancy of Head and Neck Cancer Patients in the Palliative Phase
Brief Title: Prognostic Counselling in Palliative Head and Neck Cancer (ProCoPall)
Acronym: ProCoPall
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Dutch Cancer Society (Other)
Responsible Party: Principal Investigator, Dr. Marinella P. J. Offerman, Associate Professor, Erasmus Medical Center
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 9109
Record Dates: First submitted 2024-10-25; First posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Squamous Cell Carcinoma of Head and Neck
Keywords: Palliative Care; Life expectancy; Counseling; Quality of life; Prognosis
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (No Intervention): Current general counselling on life expectancy
- Cohort 2 (Experimental): Individualized prognostic counselling on life expectancy
  Interventions: Other: Individualized prognostic counselling

INTERVENTIONS:
Other: Individualized prognostic counselling — Individualized prognostic counselling on life expectancy using the prognostic model 'OncologIQ Palliative'
  Arms: Cohort 2

SUMMARY:
The investigators test the effect of providing individualized prognostic information on life-expectancy to head and neck cancer patients in the palliative phase.

DETAILED DESCRIPTION:
In this prospective sequential cohort study, the investigators aim to include 160 patients with a palliative diagnosis of head and neck squamous cell carcinoma, divided into two cohorts. In cohort 1, patients will receive general prognostic counselling, while in cohort 2, patients will receive individualized prognostic counselling using the recently developed prognostic model 'OncologIQ Palliative'. Cohort 2 will commence after completion of cohort 1. The primary outcome will be decisional conflict and satisfaction with the decision-making process and proactive care planning. Additionally, we will assess whether patients undergo palliative treatment and, if so, the type of treatment received. We will also evaluate overall survival, the incidence of palliative sedation or euthanasia, and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received a palliative diagnosis of a squamous cell carcinoma of the oral cavity, oropharynx, nasopharynx, hypopharynx, supraglottic larynx, glottis larynx and unknown primary.

Exclusion Criteria:

* Illiterate patients
* Insufficient knowledge of Dutch language
* Incompetent (due to i.e. mental state) to consider their own treatment choice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict | 2 weeks
  Decisional conflict (DC) will be assessed using the Decisional Conflict Scale (DCS) questionnaire, reported two weeks after the consultation in which the palliative diagnosis is shared. The overall score can range from 0 (no DC) to 100 (extremely high DC). A score of ≥25 is considered the cutoff for clinically significant decisional conflict.
Satisfaction with decision making process and proactive care planning | 3-4 weeks
  To measure satisfaction with decision making process and proactive care planning, including end-of-life discussions on preferred place of death and wishes for palliative sedation and euthanasia we will conduct interviews among patients after counselling with OncologIQ Palliative

SECONDARY OUTCOMES:
Treatment | At the end of the study
  The amount and type of treatment(s) the patient receives in the palliative phase
Survival | Through study completion, up to 2 years
  Overall survival from the start of the palliative trajectory
Quality of Life Score | Baseline and every 6-8 weeks
  Quality of life will be assessed using the validated questionnaire EORTC QLQ-C15-PAL at baseline and at regular intervals throughout the study period.
  It consists of 15 questions, assessing 10 domains. All questions are scored on a 4-point scale, ranging from 1 (not at all) to 4 (very much). A higher score indicates a better QoL for the domains of emotional functioning, physical functioning, and global health status. In contrast, for the remaining domains, lower scores indicate better QoL.
Palliative sedation and Euthanasia | Through study completion, up to 2 years
  The incidence of palliative sedation and euthanasia

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van den Besselaar BN, Sewnaik A, Dorr MC, Hoesseini A, Hardillo JA, Baatenburg de Jong RJ, Offerman MPJ. A study protocol for individualized prognostic counselling in the palliative phase. BMC Palliat Care. 2025 Jan 10;24(1):9. doi: 10.1186/s12904-025-01647-z. PMID 39794711